CLINICAL TRIAL: NCT01415752
Title: Intergroup Randomized Phase 2 Four Arm Study In Patients ≥ 60 With Previously Untreated Mantle Cell Lymphoma Of Therapy With: Arm A = Rituximab+ Bendamustine Followed By Rituximab Consolidation (RB → R); Arm B = Rituximab + Bendamustine + Bortezomib Followed By Rituximab Consolidation (RBV→ R), Arm C = Rituximab + Bendamustine Followed By Lenalidomide + Rituximab Consolidation (RB → LR) or Arm D = Rituximab + Bendamustine + Bortezomib Followed By Lenalidomide + Rituximab Consolidation (RBV → LR)
Brief Title: Rituximab, Bendamustine Hydrochloride, and Bortezomib Followed by Rituximab and Lenalidomide in Treating Older Patients With Previously Untreated Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1411; NCI-2011-02980 (Other: NCI); CDR0000707057 (Other: NCI)
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma; Mantle Cell Lymphoma
Keywords: Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Induction: (A) Bendamustine + Rituximab then Maintenance: (E) Rituximab (Experimental): Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustine
- Induction: (B) Bendamustine + Rituximab + Bortezomib then Maintenance: (F) Rituximab (Experimental): Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustine; Drug: bortezomib
- Induction: (C) Bendamustine + Rituximab then Maintenance: (G) Lenalidomide + Rituximab (Experimental): Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustine; Drug: lenalidomide
- Induction: (D) Bendamustine + Rituximab + Bortezomib then Maintenance: (H) Lenalidomide + Rituximab (Experimental): Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustine; Drug: bortezomib; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; Chimeric anti-CD20 monoclonal antibody; Rituxan
Drug: Bendamustine — Given IV
  Other Names: bendamustine hydrochloride; CEP-18083; TREANDA; BENDEKA
Drug: bortezomib — Given IV or SC
  Other Names: MLN341; LDP-341; Velcade®
  Arms: Induction: (B) Bendamustine + Rituximab + Bortezomib then Maintenance: (F) Rituximab; Induction: (D) Bendamustine + Rituximab + Bortezomib then Maintenance: (H) Lenalidomide + Rituximab
Drug: lenalidomide — Given PO
  Other Names: IMiDTM compound CC-5013; Revlimid®
  Arms: Induction: (C) Bendamustine + Rituximab then Maintenance: (G) Lenalidomide + Rituximab; Induction: (D) Bendamustine + Rituximab + Bortezomib then Maintenance: (H) Lenalidomide + Rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and help kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as bendamustine hydrochloride, also work in different ways to kill cancer cells or stop them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stop the growth of mantle cell lymphoma by blocking blood flow to the cancer. It is not yet known whether giving rituximab together with bendamustine and bortezomib is more effective than rituximab and bendamustine, followed by rituximab alone or with lenalidomide in treating mantle cell lymphoma.

PURPOSE: This randomized phase II trial studies rituximab, bortezomib, bendamustine, and lenalidomide in treating previously untreated older patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the addition of bortezomib (RBV) to an induction regimen of rituximab-bendamustine (RB) improves progression-free survival (PFS) compared to RB alone in patients with previously untreated mantle cell lymphoma.
* To determine whether the addition of lenalidomide to a consolidation regimen of rituximab following an induction regimen of RB or RBV improves PFS compared to consolidation rituximab alone in this patient population.

Secondary

* To determine whether the addition of bortezomib to induction therapy improves the positron emission tomography (PET)-documented complete response (CR) rate compared to RB alone.
* To determine the objective response rate (ORR) for RB and RBV.
* Among patients who do not have PET-documented CR at the end of induction, to determine whether the addition of lenalidomide to consolidation therapy improves CR and ORR compared with rituximab alone.
* To determine overall survival (OS) in the treatment arms.
* To determine safety, with attention to the addition of bortezomib in the induction regimen and lenalidomide-rituximab (LR) as consolidation therapy.

Laboratory

* To collect paraffin-embedded tissue for creation of tissue microarray.
* To collect and bank serum and blood mononuclear cells for future studies.
* To collect formalin-fixed paraffin-embedded (FFPE) tissue to analyze potential prognostic factors (Ki-67 proliferation index by immunohistochemistry and correlation with proposed 5-gene set of proliferation markers analyzed by RNA PCR; SOX 11 expression by immunohistochemistry; and Micro-RNA levels by microarray).

Quality of Life

* Using patient-reported outcomes data, to determine the extent and severity of neuropathy associated with the addition of bortezomib to induction treatment.
* Using patient-reported outcomes data, to determine the extent and severity of fatigue associated with the addition of lenalidomide to consolidation treatment.
* To evaluate the effects of the addition of bortezomib and lenalidomide on patient-reported health-related quality of life.
* To evaluate the effects of bortezomib-related neuropathy on patient-reported health-related quality of life.
* To evaluate the response of lymphoma-specific symptoms to treatment.
* Using longitudinal patient-reported outcomes data, to describe the trajectory of lymphoma symptoms, neuropathy, fatigue, and overall health-related quality of life prior to, during, and following treatment among older adults with MCL.

Imaging

* To assess the proportion of patients up and down staging when fludeoxyglucose F 18- (FDG) PET/CT is added to standard Ann Arbor staging.
* To assess the ability of pre-treatment FDG-PET/CT (SUVmax) to predict response rate and PFS.
* Among patients with interim (post-cycle 3) FDG-PET/CT imaging, to assess the correlation of interim FDG-PET/CT imaging with response rate and PFS both during induction and consolidation therapy.
* To assess standard FDG-PET/CT metrics including SUVmax, tumor metabolic burden, total tumor burden, and association with pathology features (blastoid variant vs other, and Ki67) in the setting of MCL.
* To assess differences in overall and CR rates when using Deauville vs International Harmonization Project FDG-PET/CT interpretation criteria.
* To determine whether there is a correlation between FDG-PET/CT response and residual disease assessment by molecular and/or flow cytometric techniques.

Residual Disease Assessment by Molecular and Flow Cytometric Techniques

* To determine whether the number of malignant cells in circulation predict the number of cells in marrow.
* To determine whether the number of malignant cells in circulation/in marrow at the end of induction correlate with CR and 2-year PFS.
* To determine whether there is a higher rate of minimal residual disease (MRD) negativity among patients randomized to RBV as compared with RB, and among patients treated with LR maintenance compared with rituximab.
* To compare the two methods of MRD detection - molecular techniques and flow cytometry - as prognostic markers for outcome.

OUTLINE: This is a multicenter study. Patients are stratified according to mantle cell lymphoma International Prognostic Index risk score (low vs intermediate vs high). Patients are randomized to 1 of 4 treatment arms.

* Arm A: Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

  * Arm E: Patients receive consolidation therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm B: Patients receive induction therapy comprising bortezomib IV or subcutaneously (SC) on days 1, 4, 8, and 11 and rituximab and bendamustine hydrochloride as patients in arm A. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

  * Arm F: Patients receive consolidation therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm C: Patients receive induction therapy comprising rituximab and bendamustine hydrochloride as patients in arm A. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

  * Arm G: Patients receive consolidation therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm D: Patients receive bortezomib, rituximab, and bendamustine hydrochloride as patients in arm B. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

  * Arm H: Patients receive consolidation therapy comprising lenalidomide PO daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood and bone marrow sample collection at baseline and during treatment for correlative studies.

Patients complete the Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym), the FACT/GOG-Neurotoxicity scale (FACT/GOG-Ntx), FACT-Fatigue, and FACT-General questionnaires at baseline and periodically during study and follow up.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually for 10 years.

ELIGIBILITY:
Step 1 (Induction) Inclusion Criteria:

* Mantle Cell Lymphoma International Prognostic Index (MIPI) score must be calculated and entered in OPEN
* Histologically confirmed untreated mantle cell lymphoma (MCL), with documented cyclin D1 by immunohistochemical stains and/or t(11;14) by cytogenetics or fluorescence in situ hybridization (FISH)
* Patients must have at least one objective measurable disease parameter
* Negative pregnancy test
* Women of childbearing potential and sexually active males use an accepted and effective method of contraception
* ECOG performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mcL (1.5 x 10^9/L)
* Platelets ≥ 100,000/mcL (100 x 10^9/L)
* Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* Calculated creatinine clearance by Cockroft-Gault formula ≥ 30 mL/min
* Patient agrees that if randomized to Arms C or D, and proceeding onto Arms G or H, they must register into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist. Patients must have no medical contra-indications to, and be willing to take, DVT prophylaxis as all patients registering to the lenalidomide/rituximab Arms G and H will be required to have deep vein thrombosis (DVT) prophylaxis. Patients randomized to Arms G or H who have a history of a thrombotic vascular event will be required to have full anticoagulation, therapeutic doses of low molecular weight heparin or warfarin to maintain an INR between 2.0 - 3.0, or any other accepted full anticoagulation regimen (e.g. direct thrombin inhibitors or Factor Xa inhibitors) with appropriate monitoring for that agent. Patients on Arms G and H without a history of a thromboembolic event are required to take a daily aspirin (81 mg or 325 mg) for DVT prophylaxis. Patients who are unable to tolerate aspirin should receive low molecular weight heparin therapy or warfarin treatment or another accepted full anticoagulation regimen. Ways to minimize risk of DVT should be discussed with patients, including, but not limited to, avoiding smoking, minimizing prothrombotic hormone replacement, avoiding prolonged periods of inactivity (e.g. uninterrupted long car or plane trips).
* HIV-positive patients are not excluded but, to enroll, must meet all of the below criteria:

  * HIV is sensitive to antiretroviral therapy
  * Must be willing to take effective antiretroviral therapy, if indicated
  * CD4 count at screening >= 300 cells/mm³
  * If on antiretroviral therapy, must not be taking zidovudine or stavudine
  * Must be willing to take prophylaxis for Pneumocystis jiroveci pneumonia (PCP) during therapy and until at least 2 months following the completion of therapy or until the CD4 cells recover to over 250 cells/mm³, whichever occurs later

Step 1 (Induction) Exclusion Criteria:

* Women (sexually mature female) must not be pregnant or breast-feeding
* Evidence of prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical carcinoma, low grade prostate carcinoma (Gleason grade ≤ 6) managed with observation that has been stable for at least 6 months, or any malignancy treated with curative intent continuously disease free for >=3 years so as not to interfere with interpretation of radiographic response
* Prior therapy for MCL, except: < 2 weeks of steroid therapy for symptom control or local radiation therapy for symptom control if there is measurable disease outside the radiation portal. Patients may be on chronic steroids for non-malignant disease if on a stable dose equivalent to ≤ 20 mg prednisone per day.
* CNS involvement
* History of AIDS-defining conditions
* Grade 2 or greater peripheral neuropathy.
* NYHA Class III or IV heart failure, uncontrolled angina severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia
* Hypersensitivity to bortezomib, boron or mannitol
* A serious medical or psychiatric illness likely to interfere with study participation
* Participating in any other therapeutic clinical trial or taking any other experimental medications within 14 days prior to registration.

Step 2 (Maintenance) Inclusion Criteria:

* ECOG performance status between 0-2
* Complete response, partial response or stable disease after Step 1
* ANC >= 1000 cells/mm3 (1.0 x 10^9/L)
* Platelets >= 75,000 cells/mm3 (75 x 10^9/L)
* AST/ALT <= 2 x upper limit of normal (ULN)
* Total bilirubin <= 2 x upper limit of normal (ULN) or, if total elevated, direct bilirubin <= 2 x upper limit of normal (ULN)
* Calculated creatinine clearance by Cockroft-Gault formula >= 30 ml/min
* Patient agrees that if randomized to Arms C or D, and proceeding onto Arms G or H, they must register into the mandatory REMS program, and be willing and able to comply with the requirements of REMS.

  * Pregnancy tests must occur within 10 - 14 days and again within 24 hours prior to initiation of Cycle 1 of lenalidomide.
  * Females of childbearing potential (FCBP)* with regular or no menstruation must have a pregnancy test weekly for the first 28 days and then every 28 days while on lenalidomide therapy (including breaks in therapy); at discontinuation of lenalidomide and at Day 28 post the last dose of lenalidomide. Females with irregular menstruation must have a pregnancy test weekly for the first 28 days and then every 14 days while on lenalidomide therapy (including breaks in therapy), at discontinuation of lenalidomide and at Day 14 and Day 28 post the last dose of lenalidomide (see Appendix VI: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods).
  * Females of childbearing potential (FCBP)* must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting Cycle 1 of lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
  * A female of childbearing potential is any sexually mature female, regardless of sexual orientation of whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
  * Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study/lenaliomide: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study including interruptions in therapy; and 3) for at least 28 days after discontinuation/stopping lenalidomide. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
  * Women must agree to abstain from donating blood during study participation and for at least 28 days after discontinuation from protocol treatment.
  * Males must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from protocol treatment. All males, regardless of whether they have undergone a successful vasectomy, must agree to use a latex condom during sexual contact with a female of childbearing potential, or to practice complete abstinence from heterosexual intercourse with any female of childbearing potential during all cycles of study treatment and for at least 28 days following discontinuation of protocol treatment
  * Patients must have no medical contra-indications to, and be willing to take, DVT prophylaxis as all patients registering to the lenalidomide/rituximab Arms G and H will be required to have deep vein thrombosis (DVT) prophylaxis. Patients randomized to Arms G or H who have full anticoagulation, a history of a thrombotic vascular event will be required to have therapeutic doses of low molecular weight heparin or warfarin to maintain an INR between 2.0 - 3.0, or any other accepted full anticoagulation regimen (e.g. direct thrombin inhibitors or Factor Xa inhibitors) with appropriate monitoring for that agent. Patients on Arms G and H without a history of a thromboembolic event are required to take a daily aspirin (81 mg or 325 mg) for DVT prophylaxis. Patients who are unable to tolerate aspirin should receive low molecular weight heparin therapy or warfarin treatment or another accepted full anticoagulation regimen. Ways to minimize risk of DVT should be discussed with patients, including, but not limited to, avoiding smoking, minimizing pro-thrombotic hormone replacement, avoiding prolonged periods of inactivity (e.g. uninterrupted long car or plane trips).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2031-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Smith, MD, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (418):
- United States (416):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Baptist Cancer Institute, Jacksonville, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer, Sandpoint, Idaho
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City CCOP, Prairie Village, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center Nashua, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Hematology Oncology Associates of Central New York-Liverpool, Liverpool, New York
  - Orange Regional Medical Center, Middletown, New York
  - Mount Sinai Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology and Hematology Care Inc-Taft, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Kingsport, Kingsport, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Saint John Medical Center, Longview, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (2):
  - The Moncton Hospital, Moncton, New Brunswick
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Smith MR, Jegede OA, Martin P, Till BG, Parekh SS, Yang DT, Hsi ED, Witzig T, Dave S, Scott D, Hanson C, Kostakoglu Shields L, Abdel-Samad N, Casulo C, Bartlett NL, Caimi PF, Al Baghdadi T, Blum KA, Romer MD, Inwards DJ, Lerner RE, Wagner LI, Little RF, Friedberg JW, Leonard JP, Kahl BS. Randomized study of induction with bendamustine-rituximab +/- bortezomib and maintenance with rituximab +/- lenalidomide for MCL. Blood. 2024 Sep 5;144(10):1083-1092. doi: 10.1182/blood.2024023962. PMID 38820500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2012 to 2016, 373 patients were enrolled in this trial.
Groups:
- Induction: Bendamustine + Rituximab Then Maintenance: Rituximab: Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Rituximab: Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Induction: Bendamustine + Rituximab Then Maintenance: Lenalidomide + Rituximab: Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Lenalidomide + Rituximab: Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
Period: Induction (Step 1)
Arm/Group | Induction: Bendamustine + Rituximab Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab Then Maintenance: Lenalidomide + Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Lenalidomide + Rituximab
Started | 94 | 93 | 93 | 93
Included in the Analysis of Adverse Events | 93 | 92 | 93 | 92
Included in the Efficacy Analysis | 90 | 90 | 89 | 89
Completed | 90 | 90 | 89 | 89
Not Completed | 4 | 3 | 4 | 4
Not completed — Ineligible | 4 | 3 | 4 | 4
Period: Maintenance (Step 2)
Arm/Group | Induction: Bendamustine + Rituximab Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab Then Maintenance: Lenalidomide + Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Lenalidomide + Rituximab
Started | 75 | 68 | 76 | 74
Included in the Analysis of Adverse Events | 74 | 68 | 73 | 73
Included in the Efficacy Analysis | 70 | 66 | 69 | 71
Completed | 48 | 43 | 43 | 52
Not Completed | 27 | 25 | 33 | 22
Not completed — Lack of Efficacy | 12 | 10 | 8 | 3
Not completed — Adverse Event | 3 | 4 | 9 | 6
Not completed — Death | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 3
Not completed — Alternative therapy | 0 | 1 | 0 | 0
Not completed — Other reasons | 3 | 6 | 4 | 6
Not completed — Did not receive treatment | 1 | 0 | 2 | 1
Not completed — ineligible | 1 | 1 | 1 | 0
Not completed — Missing | 4 | 1 | 4 | 3

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction: Bendamustine + Rituximab Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Rituximab | Induction: Bendamustine + Rituximab Then Maintenance: Lenalidomide + Rituximab | Induction: Bendamustine + Rituximab + Bortezomib Then Maintenance: Lenalidomide + Rituximab | Total
Number analyzed (Participants) | 94 | 93 | 93 | 93 | 373
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 85] | 69 [43 to 87] | 68 [47 to 90] | 66 [42 to 83] | 67 [42 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 25 | 21 | 98
  Male | 68 | 67 | 68 | 72 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 1 | 7
  Not Hispanic or Latino | 89 | 90 | 88 | 91 | 358
  Unknown or Not Reported | 4 | 1 | 2 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 2 | 0 | 4 | 9
  White | 86 | 88 | 85 | 84 | 343
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 0 | 4 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) for Induction Phase
Description: PFS is defined as time from randomization to lymphoma progression or death. Progression is defined as:
  * Appearance of any new lesion >1.5 cm in any axis during or at the end of therapy
  * >=50% increase from nadir in the sum of products of the diameters (SPD) of any previously involved nodes or extranodal masses, or in a single involved node or extranodal mass, or the size of other lesions.
  * >=50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
  * Lesions should be PET positive if observed in a typical FDG-avid lymphoma or the lesion was PET positive before therapy unless the lesion is too small to be detected with current PET systems
Time Frame: Assessed at baseline, every 3 months for 2.5 years, every 6 months up to 10 years from end of treatment, and then annually up to 10 years and 6 months
Population: Eligible and treated patients at Step 1 (induction)
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Induction: Bendamustine + Rituximab (RB; Arms A + C): Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
- Induction: Bendamustine + Rituximab + Bortezomib (RBV; Arms B + D): Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
Arm/Group | Induction: Bendamustine + Rituximab (RB; Arms A + C) | Induction: Bendamustine + Rituximab + Bortezomib (RBV; Arms B + D)
Number analyzed (Participants) | 179 | 179
years | 5.5 [4.5 to 6.6] | 6.4 [4.8 to 7.7]
Statistical Analysis 1: Comparison: Induction: Bendamustine + Rituximab (RB; Arms A + C) vs Induction: Bendamustine + Rituximab + Bortezomib (RBV; Arms B + D); Test type: Superiority; p = 0.25, Log Rank — one-sided stratified log-rank test; one-sided stratified log-rank test

2. Primary Outcome: Progression-free Survival (PFS) for Maintenance Phase (Step 2)
Description: PFS is defined as time from Step 2 registration to lymphoma progression or death. Progression is defined as:
  * Appearance of any new lesion >1.5 cm in any axis during or at the end of therapy
  * >=50% increase from nadir in the sum of products of the diameters (SPD) of any previously involved nodes or extranodal masses, or in a single involved node or extranodal mass, or the size of other lesions.
  * >=50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
  * Lesions should be PET positive if observed in a typical FDG-avid lymphoma or the lesion was PET positive before therapy unless the lesion is too small to be detected with current PET systems
Time Frame: Assessed at registration to step 2, cycles 6, 12, 18, treatment completion, then every 3 months for 2.5 years, every 6 months up to 10 years from end of treatment, and then annually up to 10 years and 6 months
Population: Eligible and treated patients at Step 2 (maintenance)
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Maintenance: Rituximab (R; Arms E + F): Patients receive maintenance therapy comprising rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Maintenance: Lenalidomide + Rituximab (LR; Arms G + H): Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Maintenance: Rituximab (R; Arms E + F) | Maintenance: Lenalidomide + Rituximab (LR; Arms G + H)
Number analyzed (Participants) | 136 | 140
years | 5.9 [5.0 to 8.2] | 7.2 [5.5 to 7.8]
Statistical Analysis 1: Comparison: Maintenance: Rituximab (R; Arms E + F) vs Maintenance: Lenalidomide + Rituximab (LR; Arms G + H); Test type: Superiority; p = 0.178, Log Rank — one-sided stratified log-rank test; one-sided stratified log-rank test

3. Secondary Outcome: Objective Response for Induction Phase (Step 1)
Description: Objective response is defined as either complete response (CR) or partial response (PR).
  CR is defined as disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy.
  PR is defined as:
  * ≥ 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or extranodal masses
  * No increase in the size of other nodes, liver or spleen.
  * Bone marrow assessment is irrelevant for determination of a PR if the sample was positive prior to treatment. However, if positive, the cell type should be specified, e.g. large-cell lymphoma or small cleaved cell lymphoma.
  * No new sites of disease.
  * Patients who achieve a CR but have persistent morphologic bone marrow involvement will be considered partial responders.
  * When the bone marrow was involved before therapy and a clinical CR was achieved, but with no bone marrow assessment after treatment, patients are considered partial responders.
Time Frame: Assessed at baseline and 24 weeks (end of cycle 6)
Population: Eligible and treated patients at Step 1 (induction)
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Bendamustine + Rituximab (RB; Arms A + C) | Induction: Bendamustine + Rituximab + Bortezomib (RBV; Arms B + D)
Number analyzed (Participants) | 179 | 179
Participants
  Objective response | 158 | 158
  No objective response | 21 | 21

4. Secondary Outcome: PET-documented Complete Response for Induction Phase (Step 1)
Description: Complete response is defined as disappearance of all detectable clinical evidence of disease.
Time Frame: Assessed at baseline and 24 weeks (end of cycle 6)
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS) Rate at 5 Years Since Maintenance (Step 2)
Description: OS is defined as the time from registration of Step 2 (maintenance) until death from any cause or last know alive. The Kaplan-Meier estimate of 5-year OS rate is reported.
Time Frame: Assessed every 3 months for 2.5 years, every 6 months for years 2.5-5
Population: Eligible and treated patients for the maintenance phase (Step 2)
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- Induction: (A) Bendamustine + Rituximab Then Maintenance: (E) Rituximab: Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustine: Given IV
- Induction: (B) Bendamustine + Rituximab + Bortezomib Then Maintenance: (F) Rituximab: Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustine: Given IV
  bortezomib: Given IV or SC
- Induction: (C) Bendamustine + Rituximab Then Maintenance: (G) Lenalidomide + Rituximab: Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustine: Given IV
  lenalidomide: Given PO
- Induction: (D) Bendamustine + Rituximab + Bortezomib Then Maintenance: (H) Lenalidomide + Rituximab: Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
  Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustine: Given IV
  bortezomib: Given IV or SC
  lenalidomide: Given PO
Arm/Group | Induction: (A) Bendamustine + Rituximab Then Maintenance: (E) Rituximab | Induction: (B) Bendamustine + Rituximab + Bortezomib Then Maintenance: (F) Rituximab | Induction: (C) Bendamustine + Rituximab Then Maintenance: (G) Lenalidomide + Rituximab | Induction: (D) Bendamustine + Rituximab + Bortezomib Then Maintenance: (H) Lenalidomide + Rituximab
Number analyzed (Participants) | 70 | 66 | 69 | 71
Proportion of participants | 0.866 [0.758 to 0.928] | 0.828 [0.711 to 0.901] | 0.727 [0.602 to 0.819] | 0.853 [0.743 to 0.918]

6. Secondary Outcome: Objective Response for Maintenance (Step 2) Among Patients Without PET-documented CR at the End of Induction
Description: as for outcome 3
Time Frame: Assessed at baseline and every 4 months for 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: To Collect Paraffin Embedded Tissue for Creation of Tissue Microarray
Description: Collection of paraffin embedded tissue for creation of tissue microarray
Time Frame: Assessed at baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: To Collect and Bank Serum and Blood Mononuclear Cells for Future Studies
Description: Collecting and banking serum and blood mononuclear cells for future studies
Time Frame: Assessed at baseline, end of cycle 3, end of cycle 6, every 4 months during first year of maintenance, every 6 months during 2nd year of maintenance, and 12 months after completion of maintenance
Reporting Status: Not Posted

9. Other Pre Specified Outcome: To Collect Formalin Fixed Paraffin Embedded (FFPE) Tissue to Analyze Potential Prognostic Factors
Description: Collection of formalin fixed paraffin embedded (FFPE) tissue for future analysis of potential prognostic factors
Time Frame: Assessed at baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-Ntx Subscale) Score
Description: FACT/GOG-Ntx subscale has 11 items and the score ranges from 0 to 44. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Scale Score
Description: FACIT-Fatigue scale has 14 items and the score ranges from 0 to 56. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) Score
Description: FACT-G subscale has 27 items and the score ranges from 0 to 108. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: To Evaluate the Effects of Bortezomib-related Neuropathy (FACT/GOG-Ntx Subscale Score) on Patient Reported Health-related Quality of Life (FACT-G Score).
Description: FACT/GOG-Ntx subscale has 11 items and the score ranges from 0 to 44. FACT-G has 27 items and the score ranges from 0 to 108. The higher the score, the better the quality of life for both scales.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lymphoma) Subscale Score
Description: FACT-Lymphoma has 15 items and the score ranges from 0 to 60. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

15. Other Pre Specified Outcome: To Evaluate the Response of Lymphoma-specific Symptoms to Treatment.
Description: FACT-Lymphoma has 15 items and the score ranges from 0 to 60. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

16. Other Pre Specified Outcome: The Trajectory of Overall Health-related Quality of Life
Description: The overall health-related quality of life is evaluated using FACT-G. FACT-G subscale has 27 items and the score ranges from 0 to 108. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline, 6, 12, 30, 36, 48 and 60 months
Reporting Status: Not Posted

17. Other Pre Specified Outcome: To Assess the Proportion of Patients up and Down Staging When FDGPET/CT is Added to Standard Ann Arbor Staging.
Description: Assessment of the proportion of patients up and down staging when FDGPET/CT is added to standard Ann Arbor staging will be performed.
Time Frame: Assessed at baseline and every 4 months for 2 years and every 6 months for years 3-10 and then annually up to 15 years
Reporting Status: Not Posted

18. Other Pre Specified Outcome: To Assess the Ability of Pre-treatment FDG-PET/CT Semi Quantitative Parameters Including SUVmax and Metabolic Measurements to Predict Response Rate and PFS.
Description: To assess the ability of pre-treatment FDG-PET/CT semi quantitative parameters including SUVmax and metabolic measurements to predict response rate and PFS.
Time Frame: Assessed at baseline and every 4 months for 2 years and every 6 months for years 3-10 and then annually up to 15 years
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Assessment of the Correlation of Interim FDG-PET/CT Imaging With Response Rate and PFS Both During Induction and Consolidation Therapy
Description: Among patients with interim FDG-PET/CT imaging, to assess the correlation of interim FDG-PET/CT imaging with response rate and PFS both during induction and consolidation therapy.
Time Frame: Assessed at baseline and every 4 months for 2 years and every 6 months for years 3-10 and then annually up to 15 years
Reporting Status: Not Posted

20. Other Pre Specified Outcome: To Assess Standard FDG-PET/CT Metrics and Association With Pathology Features
Description: To assess standard FDG-PET/CT metrics including SUVmax, tumor metabolic burden, total tumor burden, and association with pathology features (blastoid variant vs. other, and Ki67) in the setting of MCL.
Time Frame: Assessed at baseline and every 4 months for 2 years and every 6 months for years 3-10 and then annually up to 15 years
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Difference in Overall Response Rates Between Deauville and International Harmonization Project FDG-PET/CT Interpretation Criteria
Description: To assess differences in overall and complete response rates when using Deauville vs. International Harmonization Project FDG-PET/CT interpretation criteria.
Time Frame: Assessed at baseline and every 4 months for 2 years
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Correlation Between FDG-PET/CT Response and Residual Disease
Description: To determine whether there is a correlation between FDG-PET/CT response and residual disease assessment by molecular and/or flow cytometric techniques
Time Frame: Assessed at baseline and every 4 months for 2 years and every 6 months for years 3-10 and then annually up to 15 years
Reporting Status: Not Posted

23. Other Pre Specified Outcome: To Determine Whether the Number of Malignant Cells in Circulation Predict the Number of Cells in Marrow
Description: To determine whether the number of malignant cells in circulation predict the number of cells in marrow
Time Frame: Assessed at baseline and end of cycle 6
Reporting Status: Not Posted

24. Other Pre Specified Outcome: The Association Between the Number of Malignant Cells in Circulation or Marrow at the End of Induction and Clinical Outcomes
Description: To determine whether the number of malignant cells in circulation/in marrow at the end of induction correlate with CR and 2 year PFS
Time Frame: Assessed at baseline and every 4 months for 2 years
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Proportion of Patients With Minimal Residual Disease (MRD)
Description: Minimal residual disease (MRD) will be evaluated using blood samples and bone marrow samples collected on this study.
Time Frame: Assessed at baseline, end of cycles 3 and 6, every 4 months during 1st year of maintenance, every 6 months during 2nd year of maintenance and 12 months after completion of maintenance
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Difference in MRD Levels by Molecular Techniques and Flow Cytometry
Description: MRD levels will be evaluated using two different methods, molecular techniques and flow cytometry. The difference in MRD levels between the two methods will be assessed.
Time Frame: as for outcome 25
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 10 years and 6 months for Arms A, B, C and D, and up to 10 years for Arms E, F, G and H.
Description: Patients who received treatment were included in the analysis of adverse events. All patients enrolled on this study were included in the analysis of all-cause mortality.
Groups:
- Induction: Bendamustine + Rituximab (Arm A); Induction: Bendamustine + Rituximab (Arm C): Patients receive induction therapy comprising rituximab IV on day 1 and bendamustine hydrochloride IV over 60 minutes on days 1-2. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
- Induction: Bendamustine + Rituximab + Bortezomib (Arm B); Induction: Bendamustine + Rituximab + Bortezomib (Arm D): Patients receive induction therapy comprising rituximab IV on day 1, bendamustine hydrochloride IV over 60 minutes on days 1-2 and bortezomib IV subcutaneously (SC) on days 1 and 8. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to maintenance treatment.
- Maintenance: Rituximab (Arm E); Maintenance: Rituximab (Arm F): Patients receive maintenance therapy comprising rituximab IV on day 1. Courses repeat every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Maintenance: Lenalidomide + Rituximab (Arm G); Maintenance: Lenalidomide + Rituximab (Arm H): Patients receive maintenance therapy comprising lenalidomide orally (PO) daily on days 1-21 every 4 weeks and rituximab IV every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Induction: Bendamustine + Rituximab (Arm A) | Induction: Bendamustine + Rituximab + Bortezomib (Arm B) | Induction: Bendamustine + Rituximab (Arm C) | Induction: Bendamustine + Rituximab + Bortezomib (Arm D) | Maintenance: Rituximab (Arm E) | Maintenance: Rituximab (Arm F) | Maintenance: Lenalidomide + Rituximab (Arm G) | Maintenance: Lenalidomide + Rituximab (Arm H)
All-Cause Mortality (participants affected / at risk) | 11/94 | 16/93 | 11/93 | 11/93 | 22/75 | 20/68 | 26/76 | 17/74
Serious Adverse Events (participants affected / at risk) | 75/93 | 80/92 | 70/93 | 83/92 | 50/74 | 41/68 | 62/73 | 65/73
Other Adverse Events (participants affected / at risk) | 92/93 | 88/92 | 93/93 | 92/92 | 71/74 | 64/68 | 73/73 | 73/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Bendamustine + Rituximab (Arm A) (N=93) | Induction: Bendamustine + Rituximab + Bortezomib (Arm B) (N=92) | Induction: Bendamustine + Rituximab (Arm C) (N=93) | Induction: Bendamustine + Rituximab + Bortezomib (Arm D) (N=92) | Maintenance: Rituximab (Arm E) (N=74) | Maintenance: Rituximab (Arm F) (N=68) | Maintenance: Lenalidomide + Rituximab (Arm G) (N=73) | Maintenance: Lenalidomide + Rituximab (Arm H) (N=73)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 4 | 5 | 1 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 4 | 4 | 1 | 4 | 5 | 5
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Edema limbs (General disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 3 | 0 | 1 | 3 | 5
Fever (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 6 | 2 | 5 | 0 | 0 | 3 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 4
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 2 | 0 | 2 | 2 | 3 | 1 | 5 | 7
Sepsis (Infections and infestations) | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 3 | 0 | 2 | 2 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INR increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 55 | 58 | 59 | 69 | 38 | 35 | 36 | 48
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 21 | 24 | 18 | 28 | 16 | 12 | 44 | 42
Platelet count decreased (Investigations) | 6 | 10 | 10 | 8 | 0 | 1 | 2 | 2
Weight gain (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
White blood cell decreased (Investigations) | 14 | 19 | 14 | 23 | 11 | 9 | 31 | 29
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0 | 3 | 0 | 1 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 7 | 3 | 3 | 3 | 3 | 2 | 3
Hypotension (Vascular disorders) | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Vascular disorders - Other, specify (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction: Bendamustine + Rituximab (Arm A) (N=93) | Induction: Bendamustine + Rituximab + Bortezomib (Arm B) (N=92) | Induction: Bendamustine + Rituximab (Arm C) (N=93) | Induction: Bendamustine + Rituximab + Bortezomib (Arm D) (N=92) | Maintenance: Rituximab (Arm E) (N=74) | Maintenance: Rituximab (Arm F) (N=68) | Maintenance: Lenalidomide + Rituximab (Arm G) (N=73) | Maintenance: Lenalidomide + Rituximab (Arm H) (N=73)
Anemia (Blood and lymphatic system disorders) | 61 | 54 | 61 | 57 | 40 | 37 | 53 | 57
Edema limbs (General disorders) | 11 | 14 | 15 | 14 | 5 | 10 | 11 | 12
Fatigue (General disorders) | 67 | 63 | 70 | 72 | 47 | 36 | 56 | 53
Fever (General disorders) | 13 | 23 | 15 | 12 | 7 | 6 | 9 | 6
Infusion related reaction (General disorders) | 13 | 14 | 12 | 5 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 9 | 6 | 7 | 5 | 3 | 16 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 6 | 0 | 1 | 5 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 26 | 24 | 22 | 5 | 3 | 28 | 25
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 2
Constipation (Gastrointestinal disorders) | 30 | 36 | 35 | 40 | 5 | 6 | 29 | 20
Diarrhea (Gastrointestinal disorders) | 16 | 34 | 19 | 26 | 7 | 9 | 35 | 31
Dyspepsia (Gastrointestinal disorders) | 9 | 9 | 9 | 7 | 4 | 1 | 5 | 4
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 41 | 48 | 40 | 51 | 10 | 8 | 20 | 14
Vomiting (Gastrointestinal disorders) | 4 | 17 | 7 | 16 | 2 | 2 | 5 | 4
Allergic reaction (Immune system disorders) | 10 | 15 | 16 | 11 | 2 | 0 | 5 | 5
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 6 | 6
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 7 | 5 | 12 | 7
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 5
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 4
Lymphocyte count decreased (Investigations) | 51 | 51 | 59 | 63 | 56 | 45 | 55 | 62
Neutrophil count decreased (Investigations) | 40 | 43 | 43 | 39 | 28 | 28 | 58 | 54
Platelet count decreased (Investigations) | 55 | 54 | 51 | 52 | 28 | 28 | 38 | 41
Weight loss (Investigations) | 10 | 14 | 14 | 17 | 2 | 7 | 6 | 9
White blood cell decreased (Investigations) | 68 | 60 | 67 | 63 | 50 | 44 | 62 | 61
Anorexia (Metabolism and nutrition disorders) | 19 | 25 | 22 | 25 | 3 | 6 | 11 | 14
Hyponatremia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 18 | 11 | 17 | 7 | 16 | 16 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2 | 4 | 3 | 3 | 7 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4
Hypertension (Vascular disorders) | 7 | 5 | 6 | 6 | 12 | 4 | 6 | 6
Hypotension (Vascular disorders) | 5 | 6 | 9 | 8 | 2 | 1 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT01415752/Prot_SAP_000.pdf